CLINICAL TRIAL: NCT05198843
Title: Phase Ib/II Study of EPA-Based EphA2 Targeted Therapy for Patients With Metastatic Triple-Negative Inflammatory Breast Cancer
Brief Title: Testing an Omega-3 Fatty Acid-Based Anti-Cancer Therapy for Patients With Triple-Negative Inflammatory Breast Cancer That Has Spread to Other Parts of the Body
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Other - Poor accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-00004; NCI-2022-00004 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10480 (Other: University of Texas MD Anderson Cancer Center LAO); 10480 (Other: CTEP); UM1CA186688 (NIH); 2022-0246 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2022-01-19; First posted 2022-01-20 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Triple-Negative Breast Inflammatory Carcinoma
MeSH Terms: interventions — Dasatinib; eicosapentaenoic acid ethyl ester; eicosapentaenoic acid ethanolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (icosapent ethyl, dasatinib) (Experimental): Patients receive icosapent ethyl PO BID and dasatinib PO QD in each treatment cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib; Dietary Supplement: Icosapent Ethyl

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
Dietary Supplement: Icosapent Ethyl — Given PO
  Other Names: (all-Z)-5,8,11,14,17-Eicosapentaenoic Acid Ethyl Ester; AMR 101; AMR101; Cis-Eicosapentaenoic Acid Ethyl Ester; Ethyl Icosapentate; Vascepa

SUMMARY:
This phase Ib/II tests the safety, side effects, and best dose of icosapent ethyl in combination with dasatinib and whether they work to shrink tumors in patients with triple-negative inflammatory breast cancer that has spread to other places in the body (metastatic). Triple-negative inflammatory breast cancer is a type of inflammatory breast cancer in which the tumor cells do not have estrogen receptors, progesterone receptors, or large amounts of HER2/neu protein on their surface. Dasatinib is in a class of medications called tyrosine kinase inhibitors. It works by blocking the action of an abnormal protein that signals cancer cells to multiply, which may help keep cancer cells from growing. Icosapent ethyl is an omega-3 fatty acid and in a class of medications called antilipemic or lipid-regulating agents. It may decrease the amount of triglycerides and other fats made in the liver. Preclinical studies have suggested that it may reduce the growth of triple negative inflammatory breast cancer cells. Combination therapy with dasatinib and icosapent ethyl may help shrink tumors in patients with triple-negative inflammatory breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine maximum tolerated dose (MTD) of icosapent ethyl (EPA) and dasatinib in patients with metastatic triple negative inflammatory breast cancer (mTN-IBC). (Phase 1b) II. To determine the overall response rate (ORR) of EPA and dasatinib therapy in patients with mTN-IBC. (Phase 2)

SECONDARY OBJECTIVES:

I. To determine the clinical benefit rate (CBR) of EPA and dasatinib therapy in patients with mTN-IBC.

II. To determine progression-free survival (PFS) at 1 year for patients with mTN-IBC who were enrolled in the study and received EPA and dasatinib therapy.

III. To determine overall survival (OS) at 2 years for patients with mTN-IBC who were enrolled in the study and received EPA and dasatinib therapy.

IV. To determine the induction of apoptosis by EPA and dasatinib therapy.

EXPLORATORY OBJECTIVES:

I. To determine the effect of EPA and dasatinib therapy on the expression of cholesterol transporter.

II. To determine the relationship between the expression of EphA2 and the treatment response to EPA and dasatinib therapy.

III. To determine the change in Ki67 by EPA and dasatinib therapy. IV. To evaluate the change in cholesterol homeostasis and tumor membrane rigidity after EPA and dasatinib therapy.

V. To investigate the effect of EPA and dasatinib therapy on the systemic inflammation.

OUTLINE: This is a phase Ib dose-escalation study of icosapent ethyl in combination with fixed dose dasatinib, followed by a phase II study.

Patients receive icosapent ethyl orally (PO) twice daily (BID) and dasatinib PO once daily (QD) in each treatment cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of the study treatment, patients will undergo in-clinic post-treatment evaluations 1 month after their last study treatment or before starting new treatment, whichever occurs first, subsequently, patients are followed every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed mTN-IBC. TNBC is defined as:

  * < 10% estrogen receptor and progesterone receptor expression by immunohistochemistry (IHC)
  * Negative or 1+ for HER2 by IHC or negative by fluorescent in situ hybridization based on American Society of Clinical Oncology (ASCO)/College of American Pathologist (CAP) guideline
* Patients must have had or currently have a clinical diagnosis of inflammatory breast carcinoma (IBC) according to the IBC-specific clinical manifestation as determined by a multidisciplinary team
* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for the phase 2 component of the study. Measurable disease is not a criterion for eligibility for the phase 1 component of the study
* Patients must have minimum of one standard regimen exposure in a metastatic setting
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of dasatinib in combination with EPA in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status: 0-2
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Creatinine =< 1.5 x institutional ULN
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2
* Patients with distant metastasis and/or local recurrence accessible for biopsy. Metastasis to brain, lung, and bone will be considered not accessible for safety reasons
* Negative serum or urine pregnancy test for subjects with childbearing potential
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be of class 2B or better
* The effects of dasatinib on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of dasatinib administration
* Patients who are currently on bisphosphonate therapy should be able to temporarily stop bisphosphonate therapy for the duration of the study pending assessment of the need for calcium supplementation
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (3 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dasatinib or icosapent ethyl or any of its components (tocopherol, gelatin, glycerin, maltitol, and sorbitol) or other agents used in study
* Patients who have not recovered from adverse events due to prior anti-cancer therapies, (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients with known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate if they are stable, and have no evidence of new or enlarging brain metastases for at least 3 months, and are not using steroids for at least 7 days prior to trial treatment
* Patients with an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study
* Patients with a history of (non-infectious) pneumonitis that required steroids or has a current diagnosis of pneumonitis
* Patients with an active infection requiring systemic therapy
* Patients with an allergy to fish, shellfish, or omega-3 unsaturated fatty acid
* Patients who received a live vaccine within 30 days prior to the first dose of trial treatment
* Patients receiving concurrent anti-cancer therapy for metastatic disease
* Patients with uncontrolled intercurrent illness judged by the investigator to be unsafe for trial participation
* Pregnant women are excluded from this study because dasatinib is a protein tyrosine kinase (PTK) inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with dasatinib, breastfeeding should be discontinued if the mother is treated dasatinib. These potential risks may also apply to other agents used in this study
* Patients with severe hypertriglyceridemia (> 300 mg/dL-500 mg/dL) are at an unknown risk of developing pancreatitis following icosapent ethyl treatment
* Patients with diabetes who are being treated with insulin. Patients with oral medication and showing stable glycosylated hemoglobin (HbA1c) < 7% for the last three months will be eligible
* Patients who require concurrent treatment with any medications or substances that are potent inhibitors or inducers of CYP3A4 are ineligible. Efforts should be made to switch patients with gliomas or brain metastases who are taking enzyme-inducing anticonvulsant agents to other medications
* Use of antithrombotic and/or anti-platelet agents (e.g., warfarin, heparin, low molecular weight heparin, aspirin, and/or ibuprofen)
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous [IV] alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain dasatinib and icosapent ethyl tablets are excluded
* Patients may not have any clinically significant cardiovascular disease including the following:

  * Myocardial infarction or ventricular tachyarrhythmia within 6 months
  * Prolonged corrected QT (QTc) >= 480 msec (Fridericia correction)
  * Ejection fraction less than institutional normal
  * Major conduction abnormality (unless a cardiac pacemaker is present) Patients with any cardiopulmonary symptoms of unknown cause (e.g., shortness of breath, chest pain, etc.) should be evaluated by a baseline echocardiogram with or without stress test as needed in addition to electrocardiogram (EKG) to rule out QTc prolongation. The patient may be referred to a cardiologist at the discretion of the principal investigator. Patients with underlying cardiopulmonary dysfunction should be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel M. Layman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: Nov 1, 2022 to Dec 19, 2023. All recruitment was done at The University of Texas MD Anderson Cancer Center. The study was closed due to poor accrual.
Pre-assignment Details: One patient was enrolled and treated. One patient was not enrolled due to a screening failure.
Groups:
- Treatment (EPA, Dasatinib): Participants receive EPA & dasatinib in each treatment cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (EPA, Dasatinib)
Started | 1
Completed | 0
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (EPA, Dasatinib)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) for Dasatinib and Icosapent Ethyl (EPA) Combination Therapy (Phase 1b)
Description: MTD is selected based on isotonic regression. Specifically, the dose is selected as the MTD for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate. If there are ties, the higher dose level is selected when the isotonic estimate is lower than the target toxicity rate; the lower dose level is selected when the isotonic estimate is greater than or equal to the target toxicity rate.
Time Frame: Up to 2 years
Population: No efficacy data was obtained since the study was terminated early. Outcome Measure has zero total analyzed at the protocol specified restaging timepoint.
Arm/Group | Treatment (EPA, Dasatinib)
Number analyzed (Participants) | 0

2. Primary Outcome: Overall Response Rate (ORR) of Dasatinib and EPA Combination Therapy (Phase 2)
Description: the percentage of patients with a best overall response of CR (complete response) or PR (partial response)
Time Frame: Up to 2 years
Population: as for outcome 1
Arm/Group | Treatment (EPA, Dasatinib)
Number analyzed (Participants) | 0

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Will be the proportion of the patients with static disease (SD) >= 24 weeks, complete response (CR), and partial response (PR). CBR will be estimated along with a 95% exact confidence interval.
Time Frame: Up to 2 years
Population: as for outcome 1
Arm/Group | Treatment (EPA, Dasatinib)
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival
Description: Defined as the rate of patients without the progression of disease or loss to follow-up at 1 year after initiating the EPA and dasatinib combination therapy. Will be estimated using the methods of Kaplan and Meier.
Time Frame: At 1 year
Population: as for outcome 1
Arm/Group | Treatment (EPA, Dasatinib)
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Defined as the survival rate at 2 years after initiating the EPA and dasatinib combination therapy. Will be estimated using the methods of Kaplan and Meier.
Time Frame: At 2 years
Population: No efficacy data was obtained since the study was terminated early. Outcome Measure has zero total analyzed.
Arm/Group | Treatment (EPA, Dasatinib)
Number analyzed (Participants) | 0

6. Secondary Outcome: Induction of Tumor Apoptosis
Description: Tumor apoptosis will be measured by using the Luminex Apoptosis multiplex immunoassay panel (cleaved caspase-3) as well as TdT-Mediated dUTP Nick End Labeling (TUNEL) assay.
Time Frame: After cycle 2 (1 cycle = 28 days)
Population: as for outcome 1
Arm/Group | Treatment (EPA, Dasatinib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: from the start date of treatment until 30 days after the last dose of study drug, approximately 2 months.
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting.
Arm/Group | Treatment (EPA, Dasatinib)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (EPA, Dasatinib) (N=1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Weight gain (Investigations) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT05198843/Prot_SAP_000.pdf
  • Informed Consent Form: Phase I (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT05198843/ICF_001.pdf
  • Informed Consent Form: Phase II (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT05198843/ICF_002.pdf